CLINICAL TRIAL: NCT01312493
Title: Selective IMRT for Locally Advanced Head and Neck Carcinoma With Concurrent Panitumumab
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding source was terminated before enrollment of first subject
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1017
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck cancer; Phase II; Locally advanced; Panitumumab; Vectibix; Lineberger; Radiation Therapy; Intensity modulated radiation therapy (IMRT); Stage III to IVB
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Panitumumab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Panitumumab — Weekly panitumumab intravenously at a dosage of 2.5 mg/kg started one week prior to RT until RT is completed. No more than 8 treatments.
  Other Names: Vectibix
Radiation: Intensity Modulated Radiation Therapy — The dose per fraction will be 2 Gy per day. Thus, the total number of fractions will be 35. Five days a week for 7 weeks.
  Other Names: IMRT

SUMMARY:
This is a non-randomized phase II study of targeted radiotherapy (RT) administered concurrently with panitumumab in patients with locally advanced squamous carcinoma of the head and neck.

DETAILED DESCRIPTION:
This is a non-randomized phase II trial of targeted radiotherapy (RT) administered concurrently with panitumumab in patients with locally advanced squamous cell carcinoma of the head and neck. This protocol addresses patients with medical comorbidities that make them poor candidates for concurrent chemotherapy. Radiotherapy treatment will be directed at disease visible on diagnostic imaging modalities and the ipsilateral hemi-neck, sparing elective regions in the contralateral N0 hemi-neck with less than 20% chance of microscopic involvement. We explore the following hypothesis: Can acceptable locoregional disease control be obtained with less treatment-related morbidity by focusing RT on regions of gross disease, sparing regions with a low risk of harboring subclinical disease from elective RT?

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary squamous cell carcinoma arising in the oral cavity, oropharynx, hypopharynx, or larynx.
* Stage III, IVA, or IVB disease (locally advanced with no systemic metastases and without bilateral nodal disease, i.e., N2c).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 with a life expectancy >12 months.
* Patients are eligible if they have concurrent medical conditions that render them poor candidates for chemotherapy. Patients are considered to be in this group if any of the following criteria is met: Serum creatinine >1.5 mg/dl (or estimated creatinine clearance <50mL/min); Insulin dependent diabetes; SGOT, SGPT, or alkaline phosphatase >2.5 x upper limit of normal; History of significant CAD (myocardial infarction [MI], coronary artery bypass graft [CABG], coronary stents, symptomatic angina); Congestive heart failure [CHF] (LVEF <40% by echocardiogram or MUGA); nephropathy; Prior history of malignancy treated with chemotherapy; Severe chronic obstructive pulmonary disease [COPD], defined as FEV1 <1L; In the opinion of the treating physician, patient would not tolerate the administration of concurrent chemotherapy and radiation
* Age >18 years.
* The patient is medically fit to tolerate a course of definitive RT.
* The patient has adequate hematologic function defined as: absolute neutrophil count >1000/ml, hematocrit >24%, and platelet count >50,000/ml. Patients with hematocrit between 20% and 24% should undergo transfusion, and may be enrolled provided their hematocrit reaches >24%.
* The patient may have had a prior malignancy but must be disease-free for three years prior to study entry. A history of superficial non-melanoma skin cancer or in situ carcinoma of the cervix less than three years will be allowed.
* The patient must agree to use effective contraception if childbearing potential exists and continue contraception for at least 6 months following completion of the study.
* Evaluation by dental services prior to initiation of radiation therapy.
* Patient must be informed of the investigational nature of the study and sign an informed consent form.

Exclusion Criteria:

* The patient has received radiation therapy previously to the head and neck. NOTE: Previous radiotherapy for skin cancers of the head and neck are permitted if the fields do not overlap significantly.
* All gross disease has been surgically resected. NOTE: Patients who have had an excisional neck biopsy will not be eligible.
* Patient with positive contralateral neck node whether ipsilateral neck is negative or positive.
* The patient is pregnant or lactating.
* Squamous cell carcinoma arising in the nasopharynx, sinuses, salivary glands, or the primary is unknown.
* Non-squamous histologies (such as adenoid cystic or mucoepidermoid carcinoma).
* Spindle cell squamous carcinoma or mixed carcinoma/sarcoma.
* Scleroderma or active connective tissue disorder (Lupus).
* Any underlying psychological condition that would prohibit the understanding and rendering of informed consent.
* Major surgery <3 weeks prior to study entry.
* History of interstitial lung disease, e.g., pulmonary fibrosis or interstitial pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence Rate of Locally Advanced Head & Neck Cancer | 2 Years
  Imaging for recurrence via CT scan will occur at 8 weeks (+/-5 days) post-RT, and will be repeated at 6, 9, 12, and 24 months from start of treatment.

SECONDARY OUTCOMES:
Patterns of Failure | 2 Years
  Evaluate locoregional recurrences to see if they arise in regions that were spared vs. treated, and assess long-term control after salvage therapy.
Time to Relapse | first day of therapy to the first sign of progressive disease
  Imaging for recurrence via CT scan will occur at 8 weeks (+/-5 days) post-RT, and will be repeated at 6, 9, 12, and 24 months from start of treatment.
Morbidity of Treatment | From screening until 30 days after treatment
  Toxicity will be assessed according to the NCI CTCAE v4.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Hayes, MD, Principal Investigator — University of North Carolina, Chapel Hill

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Homepage — http://unclineberger.org
- See also: National Cancer Institute Homepage — http://www.cancer.gov/